CLINICAL TRIAL: NCT03321981
Title: Phase 2 Study of MCLA-128-based Combinations in Metastatic Breast Cancer (MBC): MCLA-128/Trastuzumab/Chemotherapy in HER2-positive MBC and MCLA-128/Endocrine Therapy in Estrogen Receptor Positive and Low HER2 Expression MBC
Brief Title: MCLA-128 With Trastuzumab/Chemotherapy in HER2+ and With Endocrine Therapy in ER+ and Low HER2 Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merus B.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCLA-128-CL02; 2017-002821-39 (EudraCT Number)
Record Dates: First submitted 2017-10-11; First posted 2017-10-26 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer Metastatic
Keywords: Bispecific Antibody immunoglobulin gamma-1(IgG1), Human Epidermal Growth Factor Receptor (HER)2, HER3; MCLA-128; Antibodies, bispecific; Immunologic Factors; Cytokines; combination Trastuzumab with and without Vinorelbine; zenocutuzumab
MeSH Terms: conditions — Lethal Congenital Contracture Syndrome 2 | interventions — zenocutuzumab; Trastuzumab; Vinorelbine; Fulvestrant; exemestane; Letrozole; Anastrozole

STUDY DESIGN:
Intervention Model Description: three combination treatments will be evaluated, two in Cohort 1 and one in Cohort 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 doublet (Experimental): zenocutuzumab + trastuzumab
  Interventions: Drug: Zenocutuzumab; Drug: Trastuzumab
- Cohort 1 triplet (Experimental): zenocutuzumab + trastuzumab + vinorelbine
  Interventions: Drug: Zenocutuzumab; Drug: Trastuzumab; Drug: Vinorelbine
- Cohort 2 (Experimental): zenocutuzumab + endocrine therapy
  Interventions: Drug: Zenocutuzumab; Drug: Endocrine therapy

INTERVENTIONS:
Drug: Zenocutuzumab — full length immunoglobulin gamma-1 (IgG1) bispecific antibody targeting Human Epidermal Growth Factor Receptor (HER)2 and HER3
  Other Names: MCLA-128
Drug: Trastuzumab — humanised IgG1 monoclonal antibody
  Other Names: Herceptin
  Arms: Cohort 1 doublet; Cohort 1 triplet
Drug: Vinorelbine — antineoplastic drug of vinca alkaloid family
  Other Names: Navelbine; vinorelbine tartrate
  Arms: Cohort 1 triplet
Drug: Endocrine therapy — same endocrine therapy is administered as the last line of endocrine therapy
  Other Names: fulvestrant; exemestane; letrozole; anastrazole
  Arms: Cohort 2

SUMMARY:
A Phase 2, open-label, multicenter international study will be performed to evaluate the efficacy of MCLA-128-based combinations. Three combination treatments will be evaluated, two in Cohort 1 and one in Cohort 2.

MCLA-128 (zenocutuzumab) is given in combinations in two metastatic breast cancer (MBC) populations, Human Epidermal Growth Factor Receptor (HER) 2-positive/amplified (Cohort 1) and Estrogen Receptor-positive/low HER2 expression (Cohort2).

Two combinations treatments will be evaluated in Cohort 1, the doublet and triplet. Initially zenocutuzumab is given in combination with trastuzumab in the doublet. After the safety of the doublet has been assessed in 4-6 patients, MCLA-128 is given in combination with trastuzumab and vinorelbine in the triplet, in parallel to the efficacy expansion of the doublet.

The doublet and triplet combinations are both evaluated in two steps with an initial safety run-in followed by a cohort efficacy expansion. In total up to 40 patients evaluable for efficacy are included in both the doublet and triplet.

In Cohort 2 zenocutuzumab is administered in combination with the same previous endocrine therapy on which progressive disease is radiologically documented. A total of up to 40 patients evaluable for efficacy are included in the Cohort 2.

DETAILED DESCRIPTION:
Study Design Phase 2, open-label, multicenter international study to evaluate the efficacy of MCLA-128 (zenocutuzumab)-based combinations in 2 metastatic breast cancer populations, Human Epidermal Growth Factor Receptor (HER)2-positive/amplified (Cohort 1) and estrogen receptor-positive/low-HER2 expression (Cohort 2). Three combination treatments were evaluated, 2 in Cohort 1 and 1 in Cohort 2.

Cohort 1: To be eligible, patients had to have HER2-positive/amplified metastatic breast cancer, with confirmed HER2 overexpression by Immunohistochemistry (IHC) with a score of 3+ or of 2+ combined with positive Fluorescence in Situ Hybridization (FISH), have received up to 5 lines of HER2-directed therapy in the metastatic setting, and have progressed on the most recent line per Response Evaluation Criteria In Solid Tumors Guidelines (RECIST) v1.1, and have been previously treated with trastuzumab, pertuzumab and an HER2 Antibody-Drug Conjugates (ADC) in any sequence and any setting.

Initially zenocutuzumab was administered with trastuzumab (doublet combination). Safety was reviewed by an Independent Data Monitoring Committee (IDMC). If the safety of the doublet was approved, the triplet combination of zenocutuzumab plus trastuzumab and vinorelbine was to be evaluated in parallel with the doublet combination.

The doublet and triplet Cohort 1 combinations were each evaluated in 2 steps with an initial safety run-in period in 4 to 6 patients who were reviewed by the IDMC before deciding to expand the cohort. The triplet combination go/no-go decision was made by the IDMC after evaluation of the doublet safety run-in patients (based on Adverse Avents [AEs], Serious Adverse Events [SAEs], relationship to study drug, and other clinically relevant parameters [eg, laboratory parameters], available pharmacokinetics, immunogenicity, and cytokine data). If the triplet combination was considered safe, the expansion of the doublet and triplet combinations was performed in parallel. Patients were included in the triplet or doublet in a 3:1 ratio, taking into account previous exposure to vinorelbine.

After the safety run-in, if Cohort 1 doublet and Cohort 1 triplet combination therapies were considered tolerable by the IDMC, they were each to be expanded to a total of up to 40 patients evaluable for efficacy. If the doublet combination regimen was not well tolerated, Cohort 1 was to be closed. If the triplet combination was not well tolerated but the doublet was acceptable, the doublet expansion was to be continued.

Cohort 2: To be eligible, patients had to have estrogen receptor-positive and low-HER2 expression metastatic breast cancer (IHC 1+, or IHC 2+ combined with negative FISH), and radiologic or photographic evidence of disease progression on the last line of prior endocrine therapy (administered for ≥12 weeks) that included an aromatase inhibitor (AI) or fulvestrant. Patients who had received up to 3 prior endocrine therapies in the metastatic setting and had progressed on a Cyclin-Dependent Kinase (CDK) inhibitor (in any line) were eligible.

Zenocutuzumab was administered in combination with the same previous endocrine therapy on which progressive disease was radiologically/photographically documented. Up to 40 patients evaluable for efficacy were included.

ELIGIBILITY:
Inclusion Criteria

1. Signed informed consent before initiation of any study procedures.
2. Women with histologically or cytologically confirmed breast cancer with evidence of metastatic or locally advanced disease not amenable to any local therapy with curative intent:

   2.1 Cohort 1 (zenocutuzumab + trastuzumab ± vinorelbine)
   1. Documented Human Epidermal Growth Factor Receptor (HER)2 overexpression/amplification, defined as Immunohistochemistry (IHC) 3+ positive, or IHC 2+ combined with positive Fluorescence In Situ Hybridization (FISH), based on local analysis on the most recent tumor biopsy (preferably metastatic, otherwise primary), either fresh or archival collected within 24 months before screening.
   2. Documented disease progression (by investigator assessment) on up to a maximum of 5 lines of HER2- directed therapy administered in the metastatic setting and progression on the most recent line. Trastuzumab, pertuzumab and an HER2 Antibody drug conjugates (ADC) (eg. Trastuzumab emtansine (T-DM1)) must have been previously administered in any sequence and in any setting.

   2.2 Cohort 2 (zenocutuzumab + endocrine therapy)
   1. Documented hormone receptor positive status (estrogen receptor positive and/or progesterone receptor positive), defined as ≥ 1% positive stained cells by local standards, based on local analysis on the most recent tumor biopsy.
   2. Documented low-level HER2 expression, defined as IHC HER2 1+, or IHC HER2 2+ combined with negative FISH, based on local analysis on a fresh tumor biopsy or an archival biopsy collected within 24 months before screening (preferably metastatic, otherwise primary).
   3. No more than 3 lines of prior endocrine therapy (aromatase inhibitor or fulvestrant) for metastatic disease, with radiologic or photographic evidence of disease progression on the last line, after at least 12 weeks of therapy.
   4. Progression on a cyclin-dependent kinase inhibitor.
   5. No more than 2 previous chemotherapy regimens for advanced/metastatic disease. Note: Pre/peri-menopausal women could be enrolled if amenable to be treated with the Luteinizing Hormone-Releasing Hormone (LHRH) agonist goserelin. Such patients must have commenced treatment with goserelin or an alternative LHRH agonist at least 4 weeks prior to study entry, and patients who received an alternative LHRH agonist prior to study entry must switch to goserelin for the duration of the trial.
3. At least one lesion with measurable disease as defined by Response Evaluation Criteria In Solid Tumors Guidelines (RECIST) v1.1. For Cohort 2, patients with bone-only disease were eligible, even in the absence of measurable disease. Patients with bone-only disease must have lytic or mixed lesions (lytic + sclerotic), and imaging documenting progression on the last line of hormone therapy must be available for central review.
4. Age ≥ 18 years at signature of informed consent.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy of ≥ 12 weeks, as per investigator.
7. Left ventricular ejection fraction (LVEF) ≥50% by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA).
8. Adequate organ function:

   1. Absolute neutrophil count (ANC) ≥ 1.5 X 109/L.
   2. Hemoglobin ≥ 9 g/dL.
   3. Platelets ≥ 100 x 109/L.
   4. Serum calcium within normal ranges (or corrected with supplements).
   5. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤2.5 x upper limit of normal (ULN) and total bilirubin ≤1.5 x ULN (in cases of liver involvement, ALT/AST ≤5 x ULN and total bilirubin within normal ranges was allowed).
   6. Serum creatinine ≤1.5 x ULN or creatinine clearance ≥ 60 mL/min calculated according to the Cockcroft and Gault formula or Modification of Diet in Renal Disease (MDRD) formula for patients aged >65 years (Protocol Appendix 19.2).
   7. Serum albumin >3.0 g/dL.

Exclusion Criteria

1. Central nervous system metastases that are untreated or symptomatic, or require radiation, surgery, or continued steroid therapy to control symptoms within 14 days of study entry.
2. Known leptomeningeal involvement.
3. Advanced/metastatic, symptomatic, visceral spread, with a risk of life-threatening complications in the short-term (including patients with massive uncontrolled effusions [pleural, pericardial, peritoneal], pulmonary lymphangitis, and over 50% liver involvement).
4. Participation in another interventional clinical trial or treatment with any investigational drug within 4 weeks prior to study entry.
5. Any systemic anticancer therapy within 3 weeks of the first dose of study treatment. For cytotoxic agents that have major delayed toxicity, eg, mitomycin C and nitrosoureas, or anticancer immunotherapies, a washout period of 6 weeks was required. For patients in Cohort 2, this did not apply to the most recently received hormone therapy.
6. Major surgery or radiotherapy within 3 weeks of the first dose of study treatment. Patients who received prior radiotherapy to ≥25% of bone marrow were not eligible, irrespective of when it was received.
7. Persistent grade >1 clinically-significant toxicities related to prior antineoplastic therapies (except for alopecia); stable sensory neuropathy ≤ Grade 1 National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.03 was allowed.
8. History of hypersensitivity reaction or any toxicity attributed to trastuzumab, murine proteins, or any of the excipients that warranted permanent cessation of these agents (applicable for Cohort 1 only).
9. Previous exposure to vinorelbine (applicable for Cohort 1 triplet combination only).
10. Exposure to the following cumulative anthracycline doses:

    1. Doxorubicin or liposomal doxorubicin >360 mg/m².
    2. Epirubicin >720 mg/m².
    3. Mitoxantrone >120 mg/m² and idarubicin >90 mg/m².
    4. Other anthracycline at a dose equivalent to >360 mg/m² doxorubicin
    5. For patients having received > 1 anthracycline, the cumulative dose must not exceed the equivalent of 360 mg/m² doxorubicin.
11. Chronic use of high-dose oral corticosteroid therapy (>10 mg of prednisone equivalent per day).
12. Uncontrolled hypertension (systolic >150 mmHg and/or diastolic > 00 mmHg) or unstable angina.
13. History of congestive heart failure of Class II-IV New York Heart Association (NYHA) criteria, or serious cardiac arrhythmia requiring treatment (except atrial fibrillation, paroxysmal supraventricular tachycardia).
14. History of myocardial infarction within 6 months of study entry.
15. History of prior or concomitant malignancies (other than excised non-melanoma skin cancer or cured in situ cervical carcinoma) within 3 years of study entry.
16. Current dyspnea at rest of any origin, or other diseases requiring continuous oxygen therapy.
17. Current serious illness or medical conditions including, but not limited to uncontrolled active infection, clinically significant pulmonary, metabolic, or psychiatric disorders.
18. Known human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection.
19. Pregnant or lactating women; women of childbearing potential must use effective contraception methods (patient and/or partner, eg, surgical sterilization, a reliable barrier method) prior to study entry, for the duration of study participation, and for 7 months after the last dose of zenocutuzumab/trastuzumab. See Protocol Section 8.10.
20. Patients with only non-measurable lesions other than bone metastasis (eg, pleural effusion, ascites, or other visceral locations).
21. Patients with bone-only disease with blastic-only metastasis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Wasserman, MD, Study Director — Merus B.V.
Locations (25):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - HCA Midwest Health, Kansas City, Kansas
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Grand Hôpital de Charleroi (GHdC), Charleroi
  - UZ Leuven, Leuven
- France (9):
  - Hôpital Jean Minjoz, Besançon
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmette, Marseille
  - Centre René Huguenin, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Centre Claudius Régaud, Toulouse
  - Institute Gustave Roussy, Villejuif
- Netherlands Cancer Institute NKI, Amsterdam, North Holland, Netherlands
- Portugal (3):
  - Champalimaud Clinical Centre, Lisbon
  - Hopistal San Antonio, Porto
  - Instituto Português Oncologia, Porto
- Spain (5):
  - Vall D'Hebron Institute of Oncology (VHIO), Barcelona
  - Hospital Clinic. C/Villaroel, Barcelona
  - Ramon Y Cajal Universitary Hospital, Madrid
  - Hospital Universitario 12de Octubre, Madrid
  - Instituto Valenciano de Oncologia, Valencia
- Sarah Cannon Research Institute UK, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For this study 105 were enrolled, but only 104 patients were treated. The non-treated patient was excluded prior to initiation of study treatment due to failure to meet inclusion criteria 2.2d (No progression under Cyclin-Dependent Kinase (CDK) inhibitor).
  *Abbreviations used* in this section: Progressive Disease (PD) Patient (PT) Tumor Assessment (TA)
Groups:
- Cohort 1 Doublet: zenocutuzumab + trastuzumab
  Zenocutuzumab: full length IgG1 bispecific antibody targeting HER2 and HER3
  Trastuzumab: humanised IgG1 monoclonal antibody
- Cohort 1 Triplet: zenocutuzumab + trastuzumab + vinorelbine
  Zenocutuzumab: full length IgG1 bispecific antibody targeting HER2 and HER3
  Trastuzumab: humanised IgG1 monoclonal antibody
  Vinorelbine: antineoplastic drug of vinca alkaloid family
- Cohort 2: zenocutuzumab + endocrine therapy
  Zenocutuzumab: full length IgG1 bispecific antibody targeting HER2 and HER3
  Endocrine therapy: same endocrine therapy is administered as the last line of endocrine therapy
Period: Overall Study
Arm/Group | Cohort 1 Doublet | Cohort 1 Triplet | Cohort 2
Started | 15 | 39 | 50
Completed | 0 | 0 | 0
Not Completed | 15 | 39 | 50
Not completed — Progressive Disease (PD) | 15 | 30 | 47
Not completed — Subject withdrawal of all treatment and follow-up with agreement for contact | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 2
Not completed — symptomatic deterioration | 0 | 1 | 1
Not completed — Lack of compliance | 0 | 1 | 0
Not completed — Subject withdrawal of all treatment and follow-up with disagreement for contact | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Subject withdrawal of investigational product | 0 | 1 | 0
Not completed — Treating physician decision due to lack of clinical benefit for patient | 0 | 1 | 0
Not completed — Scans showed PD 01JUL2019 (but the PT has received radiation and since TA05 the assessments are NE) | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Doublet | Cohort 1 Triplet | Cohort 2 | Total
Number analyzed (Participants) | 15 | 39 | 50 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 27 | 39 | 77
  >=65 years | 4 | 12 | 11 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (12.1) | 57 (12.0) | 57 (12.2) | 56 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 39 | 50 | 104
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 4 | 7
  Not Hispanic or Latino | 12 | 31 | 44 | 87
  Unknown or Not Reported | 3 | 5 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 9 | 22 | 46 | 77
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 14 | 4 | 23
Region of Enrollment [Number; unit: participants]
  Netherlands | 1 | 2 | 1 | 4
  Belgium | 2 | 0 | 8 | 10
  United States | 2 | 8 | 6 | 16
  United Kingdom | 0 | 1 | 2 | 3
  France | 9 | 18 | 20 | 47
  Portugal | 0 | 7 | 6 | 13
  Spain | 1 | 3 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate at 24 Weeks
Description: Clinical benefit rate (CBR) at 24 weeks per investigator assessment. CBR is the proportion of patients with confirmed Complete Response (CR) or Partial Response (PR), or Stable Disease (SD) lasting 24 weeks.
Time Frame: 24 weeks
Population: Per-protocol efficacy set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Doublet | Cohort 1 Triplet | Cohort 2
Number analyzed (Participants) | 14 | 31 | 43
Participants | 3 | 18 | 9

2. Secondary Outcome: Progression Free Survival (PFS) Per Investigator Assessment
Description: For assessment per Response Evaluation Criteria In Solid Tumors Guidelines (RECIST) v1.1, PFS is the time from the date of treatment start to the date of event defined as the first documented progression or death due to any cause.
Time Frame: Baseline, every 6 weeks until end of treatment, every 3 months thereafter up to 1 year after treatment (if not progressed at end of treatment)
Population: Per-protocol efficacy set
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort 1 Doublet | Cohort 1 Triplet | Cohort 2
Number analyzed (Participants) | 14 | 31 | 43
months | 1.41 [1.38 to 1.45] | 5.52 [4.11 to 7.16] | 2.61 [1.45 to 2.73]

3. Secondary Outcome: Progression Free Survival (PFS) Per Central Review
Description: For assessment per RECIST v1.1, PFS is the time from the date of treatment start to the date of event defined as the first documented progression or death due to any cause.
Time Frame: as for outcome 2
Population: Per-protocol efficacy set
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort 1 Doublet | Cohort 1 Triplet | Cohort 2
Number analyzed (Participants) | 14 | 31 | 43
months | 1.41 [1.38 to 1.45] | 5.59 [4.11 to 7.39] | 1.45 [1.45 to 2.73]

4. Secondary Outcome: Overall Response Rate (ORR) Per Investigator Assessment
Description: The proportion of patients with overall response of Complete Response or Partial Response based upon RECIST 1.1 (confirmed response).
Time Frame: as for outcome 2
Population: Per-protocol efficacy set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Doublet | Cohort 1 Triplet | Cohort 2
Number analyzed (Participants) | 14 | 31 | 43
Participants | 0 | 10 | 1

5. Secondary Outcome: Overall Response Rate (ORR) Per Central Review
Description: as for outcome 4
Time Frame: as for outcome 2
Population: Per-protocol efficacy set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Doublet | Cohort 1 Triplet | Cohort 2
Number analyzed (Participants) | 14 | 31 | 43
Participants | 0 | 6 | 0

6. Secondary Outcome: Duration of Response (DoR) Per Investigator Assessment
Description: DoR applies only to patients with a Best Overall Response (BOR) of confirmed CR or PR (RECIST v1.1). For RECIST v1.1, DoR is defined as the time from the date of the first documented response (CR or PR) to the date of first documented progression, or death due to any cause.
Time Frame: as for outcome 2
Population: Per-protocol efficacy set
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort 1 Doublet | Cohort 1 Triplet | Cohort 2
Number analyzed (Participants) | 0 | 10 | 1
months |  | 4.21 [2.79 to NA] — Insufficient number of participants with events. | 4.50

7. Secondary Outcome: Duration of Response (DoR) Per Central Review
Description: DoR applies only to patients with a BOR of confirmed CR or PR (RECIST v1.1). For RECIST v1.1, DOR is defined as the time from the date of the first documented response (CR or PR) to the date of first documented progression, or death due to any cause.
Time Frame: as for outcome 2
Population: Per-protocol efficacy set
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort 1 Doublet | Cohort 1 Triplet | Cohort 2
Number analyzed (Participants) | 0 | 6 | 0
months |  | 6.36 [4.17 to NA] — Insufficient number of participants with events |

8. Secondary Outcome: Overall Survival (OS)
Description: The time from treatment start until death due to any cause.
Time Frame: as for outcome 2
Population: Per-protocol efficacy set
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort 1 Doublet | Cohort 1 Triplet | Cohort 2
Number analyzed (Participants) | 14 | 31 | 43
months | 14.09 [9.63 to NA] — Insufficient number of participants with events | 27.33 [19.94 to NA] — Insufficient number of participants with events | 26.41 [17.51 to NA] — Insufficient number of participants with events

9. Secondary Outcome: Number of Patients With Adverse Events (AE's) Leading to Discontinuation of Study Drug
Description: Evaluation of number of participants with Adverse Events leading to leading to discontinuation of study drug
Time Frame: During study treatment and up to 30 days after last administration of study drug (median duration of zenocutuzumab exposure was 6.0 weeks for Cohort 1 doublet, 19.3 weeks for Cohort 1 triplet and 11.8 weeks for Cohort 2).
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Doublet | Cohort 1 Triplet | Cohort 2
Number analyzed (Participants) | 15 | 39 | 50
Participants | 0 | 1 | 3

10. Secondary Outcome: Number of Patients With AE's of Special Interest (AESI)
Description: AESIs for MCLA-128 combinations include:
  Infusion-related reactions (for any antibodies, known AESI for MCLA-128) Cardiotoxicity (anti-Human Epidermal Growth Factor Receptor (HER)2 therapy) Diarrhea (anti-HER2 therapy) Myelosuppression (vinorelbine)
Time Frame: as for outcome 9
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Doublet | Cohort 1 Triplet | Cohort 2
Number analyzed (Participants) | 15 | 39 | 50
Participants
  Cardiotoxicity (anti-HER2 therapy) | 1 | 3 | 0
  Diarrhea (anti-HER2 therapy) | 7 | 28 | 17
  Infusion-related reaction | 1 | 7 | 12
  Myelosuppression (vinorelbine) | NA — Study treatment did not include Vinorelbine | 18 | NA — Study treatment did not include Vinorelbine

11. Secondary Outcome: Anti-drug Antibodies Serum Titers
Description: Number of patients with anti-drug antibodies at baseline and on treatment
Time Frame: Pre-dose for each of cycles 1, 3 and 5, and every 4 cycles thereafter, and at the End of Treatment visit.
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Doublet | Cohort 1 Triplet | Cohort 2
Number analyzed (Participants) | 15 | 39 | 50
Participants
  Baseline, Anti-Drug Antibody (ADA)-Negative | 12 | 29 | 46
  Baseline, ADA-Positive | 3 | 9 | 3
  On-treatment, evaluable | 8 | 32 | 38
  On-treatment, ADA-Negative | 8 | 32 | 35
  On-treatment, ADA-Positive | 0 | 0 | 3
  Treatment-induced ADA | 0 | 0 | 3
  Treatment-boosted ADA | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: During study treatment and up to 30 days after last administration of study drug (median duration of zenocutuzumab exposure was 6.0 weeks for Cohort 1 doublet, 19.3 weeks for Cohort 1 triplet and 11.8 weeks for Cohort 2).
Arm/Group | Cohort 1 Doublet | Cohort 1 Triplet | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/15 | 1/39 | 1/50
Serious Adverse Events (participants affected / at risk) | 2/15 | 8/39 | 9/50
Other Adverse Events (participants affected / at risk) | 15/15 | 39/39 | 48/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Doublet (N=15) | Cohort 1 Triplet (N=39) | Cohort 2 (N=50)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (3)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Doublet (N=15) | Cohort 1 Triplet (N=39) | Cohort 2 (N=50)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 11 (27) | 1 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 17 (51) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (3) | 5 (8)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Eye allergy (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Eyelid sensory disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 9 (11) | 6 (8)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 7 (7)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 12 (15) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 7 (12) | 28 (46) | 17 (29)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal discharge discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 18 (23) | 14 (17)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Ulcerative gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 6 (7) | 4 (5)
Asthenia (General disorders) | 4 (7) | 18 (28) | 5 (6)
Axillary pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 4 (4) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 2 (2)
Fatigue (General disorders) | 5 (5) | 13 (18) | 11 (14)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 3 (3)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 3 (4) | 3 (3) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 3 (3) | 1 (1)
Pain (General disorders) | 1 (1) | 2 (2) | 3 (3)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 5 (9) | 6 (8)
Sense of oppression (General disorders) | 0 (0) | 0 (0) | 1 (1)
Temperature regulation disorder (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (4)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mastitis fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (3)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 2 (4) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (3) | 6 (9) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 1 (4) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 4 (9) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 1 (5) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Electrocardiogram QRS complex abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 7 (16) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (6) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 7 (10) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 6 (11) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 5 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3) | 4 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (8) | 3 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (3)
Amnesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 7 (7) | 3 (7)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 6 (8) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (4) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 3 (4) | 0 (0)
Emotional disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (3) | 3 (3)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Breast inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (8) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 6 (6) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 2 (3)
Hot flush (Vascular disorders) | 0 (0) | 2 (3) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (6)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication of results by PI before the first multi-center publication by Sponsor. If there is no multi-center publication within 18 months after the study has been completed, PI may publish subject to 45 days' notice to Sponsor to review, comment, identify confidential information to be deleted, and request delay of publishing for a maximum of 120 days to permit filing of patent applications. PI agrees to accept Sponsor's reasonable comments and suggestions with respect to such publications.

DOCUMENTS (2):
  • Study Protocol (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT03321981/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT03321981/SAP_001.pdf